CLINICAL TRIAL: NCT04212572
Title: Ultrasound Abnormalities of the Salivary Glands in Primary Sjögren's Syndrome
Brief Title: Ultrasound Abnormalities of the Salivary Glands in Primary Sjögren's Syndrome According to the Duration of the Disease
Acronym: MASAÏ
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: MASAI (29BRC19.0103)
Record Dates: First submitted 2019-12-19; First posted 2019-12-27 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Primary sjögren's Syndrome
Keywords: Primary sjögren's syndrome; ultrasonography; salivary glands; auto-immune disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Salivary gland ultrasonography is identified as a valuable diagnostic tool and potential criteria item for disease classification of sjögren's syndrome and evaluate evolution of parenchyma.

The investigators have to include 242 patients. The objective is to evaluate the modification of ultrasonographic abnormalities according to disease in primary Sjögren syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient ≥ 18 years
* Primary sjögren syndrome according of age to 2002 or 2016 classification criteria

Exclusion Criteria:

* Secondary sjögren syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Primary sjögren syndrome
Sampling Method: Probability Sample
Enrollment: 242 (Estimated)
Dates: Start 2019-11-20 (Actual); Primary Completion 2020-05-20 (Estimated); Study Completion 2020-05-20 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of parenchymal abdnormalities. | inclusion
  Presence or absence of parenchymal abdnormalities. Scored following a standardized fill and according to disease duration

SECONDARY OUTCOMES:
Parenchymal abnormalities according to disease activity | inclusion
  Ultrasonography parenchymal abnormalities of salivary gland

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHRU de Brest, Brest
  - CHU de LILLE, Lille
  - CHU de MONTEPELLIER, Montpellier

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning one year and ending two years following the publication
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.